CLINICAL TRIAL: NCT07271602
Title: Iparomlimab and Tuvonralimab (QL1706) Combined Chemotherapy and Quad Shot Radiotherapy in First-line Treatment of Driver Gene-negative Advanced Non-small Cell Lung Cancer: a Randomized, Controlled, Phase 2, Open-label Trial.
Brief Title: A Phase 2 Randomized, Controlled Trial of QL1706 Plus Chemotherapy and Quad Shot for Driver Gene-negative Advanced Non-small Cell Lung Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNION-LUNG-001
Record Dates: First submitted 2025-11-24; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; Immunotherapy; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL1706, chemotherapy, Quad shot radiotherapy (Experimental): QL1706 is combined with chemotherapy for 4 cycles. Starting from Cycle 1, concurrent Quad shot radiotherapy is administered (for a maximum of 3 cycles), followed by entry into the QL1706 maintenance treatment phase.
  Interventions: Radiation: Quad shot; Drug: Chemotherapy; Drug: Immune Checkpoint Inhibitors
- Chemotherapy, QL1706 (Placebo Comparator): QL1706 is combined with chemotherapy for a total of 4 cycles, with one cycle administered every 21 days; subsequent treatment proceeds to the QL1706 maintenance therapy phase.
  Interventions: Drug: Chemotherapy; Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Radiation: Quad shot — Intensity-modulated radiotherapy (IMRT) technique is adopted, and only partial lesions (as determined by the investigator) receive Quad shot radiotherapy. Only the gross tumor volume (GTV) is irradiated, with no prophylactic irradiation of lymph nodes. The irradiation dose for the planning gross tumor volume (PGTV) is 14.8 Gy in 4 fractions, administered twice daily (bid), with an interval of more than 6 hours between each irradiation. The treatment is repeated every 3 weeks for a total of 3 cycles.
  Arms: QL1706, chemotherapy, Quad shot radiotherapy
Drug: Chemotherapy — For patients with lung squamous cell carcinoma, TC regimen chemotherapy combined with QL1706 is administered on days 1, 22, 43, and 64, respectively. The specific TC chemotherapy regimen is as follows: nab-paclitaxel 260 mg/m², intravenous infusion; carboplatin at an AUC of 5, with the total dose (mg) calculated as AUC × (GFR + 25), where GFR refers to glomerular filtration rate, administered via intravenous infusion.
  For patients with lung adenocarcinoma, PC regimen chemotherapy combined with QL1706 is administered on days 1, 22, 43, and 64, respectively. The specific PC chemotherapy regimen is as follows: pemetrexed 500 mg/m², intravenous infusion; carboplatin at an AUC of 5, with the total dose (mg) calculated as AUC × (GFR + 25), where GFR refers to glomerular filtration rate, administered via intravenous infusion.
Drug: Immune Checkpoint Inhibitors — The specific treatment regimen for QL1706 is as follows: QL1706 (5 mg/kg) via intravenous infusion.

SUMMARY:
Chemotherapy combined with immunotherapy has become the first-line standard treatment regimen for metastatic non-small cell lung cancer (NSCLC). QL1706 is an antibody that can simultaneously block the CTLA-4 and PD-1. In a phase II clinical study, when QL1706 was combined with chemotherapy for first-line treatment of metastatic NSCLC, the median progression-free survival (mPFS) was 6.8 months and the objective response rate (ORR) was 45% at a median follow-up time of 12.6 months (range, 0.4-15.2 months).

Radiotherapy is one of the commonly used local treatment modalities for tumors, which has a synergistic effect with immunotherapy, can enhance the response to immunotherapy, and trigger the abscopal effect. Quad shot radiotherapy is a periodic pulsed hypofractionated radiotherapy, with a specific mode as follows: 2 fractions per day, with an interval of more than 6 hours between the two fractions, for 2 consecutive days, with a total dose of 14-14.8 Gy. This regimen can be repeated every 3-4 weeks for a total of 3 cycles, with a total treatment dose of approximately 44-48 Gy, and it can be used for palliative treatment of various advanced tumors.

This project intends to explore whether the addition of Quad shot radiotherapy to QL1706 combined with chemotherapy can improve local and systemic tumor control rates, prolong patients' PFS, and evaluate the safety of the combined therapy in treatment-naive patients with metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed age: 18-75 years;
2. Histologically or cytologically diagnosed as lung squamous cell carcinoma or lung adenocarcinoma;
3. Staged as stage IV (T1-4NxM1) according to the Union for International Cancer Control/American Joint Committee on Cancer (UICC/AJCC) Cancer Staging System (9th edition), with at least 2 evaluable lesions, including one distant metastatic lesion;
4. Driver gene-negative;
5. ECOG performance status: 0-1;
6. Normal bone marrow function: white blood cell count > 4×10⁹/L, hemoglobin concentration > 90 g/L, platelet count > 100×10⁹/L;
7. Normal liver and kidney function: total bilirubin ≤ 1.5×upper limit of normal (ULN); aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 2.5×ULN; alkaline phosphatase (ALP) ≤ 2.5×ULN; creatinine clearance ≥ 60 mL/min;
8. Normal results of thyroid function, amylase, lipase, pituitary function, inflammatory/infectious markers, myocardial enzymes, and electrocardiogram (ECG). For patients aged > 50 years with a smoking history, normal pulmonary function test results are required. For patients with abnormal ECG or a history of cardiovascular disease (that does not meet the exclusion criteria listed in item 7), additional myocardial function tests and echocardiography are required, with normal results;
9. Patients have signed the informed consent form and are willing and able to comply with follow-up, treatment, laboratory tests, and other study requirements as specified in the study schedule;
10. Female subjects of childbearing potential must agree to use reliable contraceptive methods (e.g., condoms, regularly used contraceptives as prescribed by a physician) from screening until 1 year after treatment.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen (HBsAg) with hepatitis B virus (HBV) DNA quantitation > 1×10³ copies/mL, or positive for anti-hepatitis C virus (HCV) antibody;
2. Positive for anti-HIV antibody or diagnosed with acquired immunodeficiency syndrome (AIDS);
3. Active pulmonary tuberculosis: Patients with a history of active tuberculosis within the past year, regardless of treatment status, should be excluded. Patients with a history of active tuberculosis more than 1 year ago should be excluded, except those with confirmed regular anti-tuberculosis treatment in the past;
4. Active, known, or suspected autoimmune diseases (including but not limited to uveitis, enteritis, hepatitis, pituitary disorders, nephritis, vasculitis, hyperthyroidism, hypothyroidism, and asthma requiring bronchodilators). Exceptions include type 1 diabetes mellitus, hypothyroidism requiring hormone replacement therapy, and skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia);
5. A history of interstitial lung disease or pneumonia within the past year requiring oral or intravenous steroid treatment;
6. Chronic systemic glucocorticoid therapy (dose equivalent to or exceeding 10 mg prednisone per day) or any other form of immunosuppressive therapy. Subjects receiving inhaled or topical corticosteroids are eligible;
7. Uncontrolled heart disease, such as: 1) Heart failure with NYHA class ≥ 2; 2) Unstable angina pectoris; 3) History of myocardial infarction within the past year; 4) Supraventricular or ventricular arrhythmias requiring treatment or intervention;
8. Pregnant or lactating women (pregnancy testing should be considered for sexually active women of childbearing age);
9. Previous or current malignant tumors other than adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary thyroid carcinoma;
10. Hypersensitivity to macromolecular protein preparations or any component of QL1706;
11. Active infection within 1 week requiring systemic treatment;
12. Receipt of live vaccines within 30 days prior to the first course of immunotherapy;
13. History of organ transplantation;
14. Other conditions assessed by investigators that may endanger patient safety or compliance, such as severe diseases requiring prompt treatment (including mental illnesses), significantly abnormal test results, or other psychological, family, or social high-risk factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1 year

IPD SHARING:
Plan to Share IPD: No